CLINICAL TRIAL: NCT05892978
Title: The Effect of Infrared Light Use on Pain, Fear, and Patient Satisfaction During Peripheral Intravenous Catheter (PIVC) Procedure in Oncology Patients Receiving Chemotherapy
Brief Title: The Effect of Infrared Light Use in Oncology Patients Receiving Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Hulya Yilmaz, Principal Investigator, PhD, Msc, Uludag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16/05/2023-11/42
Record Dates: First submitted 2023-05-29; First posted 2023-06-07 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Pain; Fear Needles; Satisfaction, Patient
Keywords: Near-infrared light; Transilluminator; Peripheral intravenous cannulation; Vascular access
MeSH Terms: conditions — Pain; Iatrophobia; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized controlled experimental study.
Masking Description: The intervention and measurements will carried out by the researcher (for hand manipulation standard) and the patients will discovered their own groups when intervention will applied to them. Because of the nature of the intervention, blinding will not be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vascular imaging device with the infrared light group (Experimental): The patient's vital signs, skin color and skin turgor will be evaluated and recorded in the PIVC procedure registration form. The skill duration will be measured and recorded by the researcher with a stopwatch. The selection of the necessary materials will not be added to this time, the chronometer will be started after the tourniquet is attached, and the time will end with the blood coming to the PIVC. Data obtained on PIVC placement; vein visibility, the catheter number used in the procedure, the time to identify the appropriate vein, the successful PIVC placement time, the number of attempts for successful catheter placement, the vein in which the catheter was placed, the pain and fear levels before, during and after the procedure. These data will be recorded in the data form regarding the PIVC application. Finally, patients will be asked about their level of satisfaction with the procedure at the end of the infusion.
  Interventions: Other: Vascular imaging
- Vascular access transillumination group (Experimental): The patient's vital signs, skin color and skin turgor will be evaluated and recorded in the PIVC procedure registration form. Before the tourniquet is attached before the procedure, the patient's vein visibility will be evaluated by the research nurse. The vein imaging device will be opened with transilluminator, the tourniquet will be connected, and the vein visibility will be re-evaluated by the operator. The skill duration will be measured and recorded by the researcher with a stopwatch. The selection of the necessary materials will not be added to this time, the chronometer will be started after the tourniquet is attached, and the time will end with the blood coming to the PIVC. Data obtained on PIVC placement; the pain and fear levels before, during and after the procedure. Finally, patients will be asked about their level of satisfaction with the procedure at the end of the infusion.
  Interventions: Other: Vascular imaging
- Control group (No Intervention): The patient's vital signs, skin color, and skin turgor will be evaluated and recorded in the PIVC procedure registration form. Before the tourniquet is attached before the procedure, the patient's vein visibility will be evaluated by the research nurse. Vein imaging will not be performed. No intervention will be carried out the tourniquet will be connected, and the vein visibility will be re-evaluated by the operator. The skill duration will be measured and recorded by the researcher with a stopwatch. The selection of the necessary materials will not be added to this time, the chronometer will be started after the tourniquet is attached, and the time will end with the blood coming to the PIVC. Data will obtained on PIVC placement; the pain and fear levels before, during, and after the procedure. Finally, patients will be asked about their level of satisfaction with the procedure at the end of the infusion.

INTERVENTIONS:
Other: Vascular imaging — Experimental group - Vascular imaging device with the infrared light group: Before PIVC, infrared light will be directed to the vein area and the procedure will be started after vein visibility is achieved.
  Experimental group - Vascular access transillumination group: Before PIVC, a transilluminator will be inserted to the vein area and the procedure will be started after vein visibility is achieved
  Other Names: Vascular imaging device with the infrared light group; Vascular access transillumination group
  Arms: Vascular access transillumination group; Vascular imaging device with the infrared light group

SUMMARY:
Purpose: This study will be conducted on the effect of infrared light on PIVC procedure fear, procedure pain, and patient satisfaction in oncology patients receiving chemotherapy treatment. The investigators will implement the study during the insert on PIVC; the vascular imaging device with the infrared light group; the vascular access transillumination group; and the control group.

Design: This is a prospective, randomized controlled experimental study.

DETAILED DESCRIPTION:
The population of the research will be cancer patients who applied to Bursa Uludag University Medical Faculty Hospital Oncology unit between June 2023 and July 2025. The population of the study will consist of patients who applied to the Chemotherapy Unit in Bursa Uludağ University Health Research and Application Center Hospital Oncology Polyclinic for outpatient treatment. It is aimed to reach all patients who agreed to participate in the study and who met the inclusion criteria of the study, rather than using the research sample selection method. However, this data does not show the number of patients who applied to the unit because of the repeated visits of the patients during the chemotherapy treatment process. For this reason, direct sample selection was not made in the study, and the sample calculation was made according to the number of patients registered in the unit and the results of previous research. Calculations were made using the "G.Power-3.17" program with 95% confidence, an effect size of 0.4, and a statistical test power of at least 80%. Accordingly, it was aimed to reach 126 patients, at least 42 in each group.However, since the losses will be ignored, it is aimed to reach 150 patients in total. The hypotheses of the research;

H0,1: In patients receiving chemotherapy, the vein imaging device has no effect on the successful PIVC procedure by determining the appropriate vein.

H1,1: In patients receiving chemotherapy, the vein imaging device has an effect on the successful PIVC procedure by determining the appropriate vein.

H2: Vascular imaging device has a lower value in terms of pain in the PIVC procedure in patients receiving chemotherapy.

H3: In patients receiving chemotherapy, the vascular imaging device has a lower level of fear in the PIVC procedure.

H4: In patients receiving chemotherapy, vascular imaging device is higher in terms of patient satisfaction in PIVC procedure.

Implementation of the study in the vascular imaging device with the infrared light group: The patient will be taken to the chemotherapy application chair and rested. The patient's vital signs, skin color and skin turgor will be evaluated and recorded in the PIVC procedure registration form. Since it is stated in the literature that the placement of the peripheral intravenous catheter in the unused arm is important in preventing complications, the PIVC procedure will be performed in the arm that the patient does not actively use. Before the tourniquet is attached before the procedure, the patient's vein visibility will be evaluated by the research nurse . The vein imaging device will be opened with infrared light, the tourniquet will be connected, and the vein visibility will be re-evaluated by the research nurse. As soon as the turnstile is connected, the stopwatch will be started. Then the PIVC placement process will be started with the help of the device. The skill duration will be measured and recorded by the researcher with a stopwatch. The selection of the necessary materials will not be added to this time, the chronometer will be started after the tourniquet is attached, and the time will end with the blood coming to the branule. If there is no blood, the attempt will be considered unsuccessful. In unsuccessful cases, the PIVC attempt will be repeated up to two times in each patient. All procedures will be performed by a single research nurse to ignore the operator hand manipulation difference. Data obtained on PIVC placement; Vein visibility, the catheter number used in the procedure, the time to identify the appropriate vein, the successful PIVC placement time, the number of attempts for successful catheter placement, the vein in which the catheter was placed, the pain and fear levels before, during and after the procedure. These data will be recorded in the data form regarding the PIK application. Finally, patients will be asked about their level of satisfaction with the procedure at the end of the infusion. The satisfaction levels in the form will be evaluated on a scale ranging from 0 to 10, with 0: none, 10: many, after the application. These data will be recorded in the data form on PIVC transaction satisfaction.

Implementation of the study in the vascular access transillumination group: The processes will be repeated exactly. Transilluminator will be used instead of infrared light.

Implementation of the study in the control group: The processes will be repeated exactly. No intervention will be made for vascular access.

ELIGIBILITY:
Inclusion Criteria:

* patients who have undergone chemotherapy treatment and have received their first cure,
* patients between the ages of 18 and 74,
* patients who have not allergic to any substance,
* patients who no peripheral vascular disease,
* patients who does not have a chronic disease diagnosed other than cancer,
* patients who does not use alcohol,
* patients who non-smoker,
* patients who not taking anticoagulant treatment,
* patients who no signs of infiltration and phlebitis,
* patients who have not acute trauma around the extremity, inflammation, ecchymosis, hematoma, scar tissue, edema, metal prosthesis, no paralysis,
* patients who no visible deformity and thrombocytopenia in the examination,
* patient who mastectomy has not been performed,
* patients who do not have communication problems and whose mental level is suitable to participate in the research will be taken.

Exclusion Criteria:

* patients who have under the age of 18 and over the age of 74,
* patients who will receive chemotherapy for the first time,
* patients who changing chemotherapy cure treatment,
* patients who allergic to any substance,
* patients who do not volunteer to participate in the study will not be included in the study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-06-17 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (Pain) | through study completion, an average of 1 year
  It is a one-dimensional scale used in the measurement of VAS pain. Among the one-dimensional scales used to determine the severity of pain in patients, it was determined that the VAS measures more sensitively and is more reliable. The scale consists of a 100 mm long horizontal line. On one end are the phrases "No Pain" and on the other end "Unbearable Pain" describing the most severe pain possible. The patient is asked to mark his pain on the scale.
  The length of the line from the starting point of the scale to the point marked by the patient is measured and recorded in mm. It includes minimum 0 point, maximum 100 points.

SECONDARY OUTCOMES:
Visual Analog Scale (Fear) | through study completion, an average of 1 year
  It is a one-dimensional scale used in the measurement of VAS fear. Among the one-dimensional scales used to determine the severity of fear in patients, it was determined that the VAS measures more sensitively and is more reliable. The scale consists of a 100 mm long horizontal line. On one end are the phrases "No Fear" and on the other end "Unbearable Fear" describing the most severe fear possible. The patient is asked to mark his/her fear on the scale.
  The length of the line from the starting point of the scale to the point marked by the patient is measured and recorded in mm. It includes minimum 0 point, maximum 100 points.

OTHER OUTCOMES:
Patient satisfaction | through study completion, an average of 1 year
  In this form, patients' satisfaction with the procedure will be evaluated using a visual comparison scale that can be graded from 1 to 10. It consists of questions created in line with the literature about how the nurse evaluates the patient's skills about the PIC procedure, how she evaluates your general PIC access experience, whether she sees herself as a patient with a history of DIFFICULT VASCULAR PATH, and whether the nurse who will perform PIC makes a comprehensive assessment of her veins (Eren and Çalışkan, 2021; Ramer et al., 2016). It includes minimum 0 point, maximum 10 points.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) doesn't share any other researchers. Only research team will see data on IPD. After the data collection phase is completed and turned into a publication, other researchers can access the publication.

REFERENCES:
- [Background] Ramer L, Hunt P, Ortega E, Knowlton J, Briggs R, Hirokawa S. Effect of Intravenous (IV) Assistive Device (VeinViewer) on IV Access Attempts, Procedural Time, and Patient and Nurse Satisfaction. J Pediatr Oncol Nurs. 2016 Jul;33(4):273-81. doi: 10.1177/1043454215600425. Epub 2015 Oct 28. PMID 26510643
- [Background] Fink RM, Hjort E, Wenger B, Cook PF, Cunningham M, Orf A, Pare W, Zwink J. The impact of dry versus moist heat on peripheral IV catheter insertion in a hematology-oncology outpatient population. Oncol Nurs Forum. 2009 Jul;36(4):E198-204. doi: 10.1188/09.ONF.E198-E204. PMID 19581223
- [Background] Aulagnier J, Hoc C, Mathieu E, Dreyfus JF, Fischler M, Le Guen M. Efficacy of AccuVein to facilitate peripheral intravenous placement in adults presenting to an emergency department: a randomized clinical trial. Acad Emerg Med. 2014 Aug;21(8):858-63. doi: 10.1111/acem.12437. PMID 25176152
- [Background] Chiao FB, Resta-Flarer F, Lesser J, Ng J, Ganz A, Pino-Luey D, Bennett H, Perkins C Jr, Witek B. Vein visualization: patient characteristic factors and efficacy of a new infrared vein finder technology. Br J Anaesth. 2013 Jun;110(6):966-71. doi: 10.1093/bja/aet003. Epub 2013 Feb 5. PMID 23384732
- [Background] Eren H, Caliskan N. Effect of a Vein Imaging Device and of Fist Clenching on Determination of an Appropriate Vein and on Catheter Placement Time in Patients Receiving Chemotherapy: A Randomized Controlled Trial. Cancer Nurs. 2022 Mar-Apr 01;45(2):105-112. doi: 10.1097/NCC.0000000000000931. PMID 33654007
- [Derived] Yilmaz H, Karacan Y, Macun S, Evrensel T. The effect of using vein visualization devices to facilitate peripheral intravenous cannulation on pain, fear, and patient satisfaction in adult oncology patients: a randomized controlled trial. Support Care Cancer. 2025 Nov 24;33(12):1123. doi: 10.1007/s00520-025-10187-4. PMID 41276617